CLINICAL TRIAL: NCT00550563
Title: Identification of 24-Hydroxylase Polymorphisms and Splicing Variants That Modulate Vitamin D Oxidative Metabolism and Serum Pharmacokinetics in Patients With Colorectal Cancer on Cholecalciferol Therapy
Brief Title: DNA Changes That Affect Vitamin D Metabolism in Patients With Colorectal Cancer Receiving Vitamin D Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 99207; RPCI-I-99207
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cholecalciferol; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Chromatography, High Pressure Liquid; Chemotherapy, Adjuvant; Radioimmunodetection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Cholecalciferol (Experimental): Patients receive oral cholecalciferol 2000 IU once daily for 1 year
  Interventions: Dietary Supplement: cholecalciferol; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: protein expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Genetic: western blotting; Other: high performance liquid chromatography; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: adjuvant therapy; Procedure: immunoscintigraphy

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Oral
Genetic: polymerase chain reaction — companion study
Genetic: polymorphism analysis — companion study
Genetic: protein expression analysis — companion study
Genetic: reverse transcriptase-polymerase chain reaction — companion study
Genetic: western blotting — companion study
Other: high performance liquid chromatography — companion study
Other: laboratory biomarker analysis — companion study
Other: pharmacological study — companion study
Procedure: adjuvant therapy — Additional therapy
Procedure: immunoscintigraphy — additional testing

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This clinical trial is studying changes in DNA that affect vitamin D metabolism in patients with colorectal cancer receiving vitamin D supplements.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify CYP24 single nucleotide polymorphisms (SNPs) using peripheral blood mononuclear cell genomic DNA from patients with colorectal cancer receiving cholecalciferol supplementation.
* To evaluate the effects of these CYP24 SNPs on baseline serum vitamin D_3 metabolites (25-D_3, 24,25-D_3, and 1,25-D_3), and parathyroid hormone levels (PTH).
* To evaluate the effects of these CYP24 SNPs on serum vitamin D_3 metabolites and PTH levels during cholecalciferol treatment.
* To examine CYP24 splicing, protein expression, and enzyme activity at baseline and during cholecalciferol treatment.
* To determine the relationship, if any, between serum cholecalciferol pharmacokinetic parameters and CYP24 SNPs, splicing variants, and enzyme activity.

OUTLINE: Patients receive oral cholecalciferol 2000 IU once daily for 1 year. Patients without response to vitamin D supplementation (serum 25-D_3 level < 32 ng/mL) by 6 months will have their cholecalciferol dose increased to 4000 IU once daily.

Blood is collected at baseline and on days 14, 30, 60, 90, 180, 270, and 360. Peripheral blood mononuclear cells for CYP24 genotyping, protein expression, enzyme activity, and splicing variants are analyzed by polymerase chain reaction (PCR), western blot, high performance liquid chromatography, and reverse transcriptase PCR, respectively. Serum is analyzed for vitamin D_3 metabolite levels (by radioimmunoassay), calcium (to monitor for hypercalcemia), and parathyroid hormone assays (to measure vitamin D effect).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior or current documented diagnosis of colorectal cancer

  * All stages
* 25OH-D3 level < 50 ng/mL

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 6 months
* Serum creatinine < 2.0 mg/dL
* Serum bilirubin < 2.0 mg/dL
* No prior or current hypercalcemia (defined as albumin corrected serum calcium < 10.2 mg/dL)
* No known contraindication for vitamin D supplementation
* No genitourinary stones within the past 5 years
* No severe comorbid conditions such as uncompensated heart failure or active infection

PRIOR CONCURRENT THERAPY:

* No supplemental vitamin D beyond what is provided through the study
* At least 2 months since prior vitamin D supplementation exceeding 800 International Units (IU)

  * Nondietary vitamin D supplements should not have exceeded 800 IU/day within the past 2 months

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-08; Primary Completion 2009-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Identification of CYP24 single nucleotide polymorphisms (SNPs) | Baseline, days 14, 30, 60, 90, 180, 270, 360
Effect of CYP24 SNPs on baseline serum vitamin D3 metabolites (25-D3, 24,25-D3, and 1,25-D3), and parathyroid hormone levels (PTH) | At baseline
Effect of CYP24 SNPs on serum vitamin D3 metabolites and PTH levels during cholecalciferol treatment | Baseline, days 14, 30, 60, 90, 180, 270, 360
CYP24 splicing, protein expression, and enzyme activity at baseline and during cholecalciferol treatment | Baseline, days 14, 30, 60, 90, 180, 270, 360
Relationship between serum cholecalciferol pharmacokinetic parameters and CYP24 SNPs, splicing variants, and enzyme activity | Baseline, days 14, 30, 60, 90, 180, 270, 360

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States